CLINICAL TRIAL: NCT00113828
Title: Non-Myeloablative HLA-Matched Ex-Vivo T-cell Depleted Stem Cell Transplantation for Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Thomas Spitzer, Director, Bone Marrow Transplant Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-222
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Lymphoma; Leukemia; Multiple Myeloma; Myelodysplastic Syndrome
Keywords: Non-Myeloablative; Stem Cell Transplantation; T-cell Depletion; HLA-Matched
MeSH Terms: conditions — Lymphoma; Leukemia; Multiple Myeloma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplantation (Experimental): T-cell depleted HLA-matched peripheral blood stem cell transplantation
  Interventions: Procedure: Non-myeloablative Ex-Vivo T-cell Depleted PBSC Transplant; Procedure: T-cell depleted peripheral blood stem cell transplant

INTERVENTIONS:
Procedure: Non-myeloablative Ex-Vivo T-cell Depleted PBSC Transplant — Rabbit anti-thymocyte globulin 0.5 mg/kg on transplant day-8, 2.5 mg/kg on day-7 and 3.0 mg/kg on day-6; cyclophosphamide 60 mg/kg on days-7,-6; fludarabine 25 mg/m2 on days -5, -4, -3, -2, -1.
  Non-myeloablative Ex-Vivo T-cell Depleted PBSC Transplant.
  Other Names: Cyclosporine iv beginning on transplant day -1
Procedure: T-cell depleted peripheral blood stem cell transplant — Rabbit anti-thymocyte globulin 0.5 mg/kg on transplant day-8, 2.5 mg/kg on day-7, 3.0 mg/kg on day-6; cyclophosphamide 60 mg/kg on days -7, -6; fludarabine 25 mg/m2 on days -5 through -1.
  T-cell depleted peripheral blood stem cell transplant .
  Other Names: Cyclosporine iv beginning on day -1.

SUMMARY:
The purpose of this trial is to determine if patients with hematologic diseases who have a HLA 6/6 matched related donor and are not eligible for a standard myeloablative stem cell transplant will have less severe graft versus host disease (GVHD), transplant related mortality, and less graft failure when treated with a non-myeloablative T-cell depleted stem cell transplant.

DETAILED DESCRIPTION:
Our prior experience in the lab and in clinical trials with non-myeloablative HLA-matched and mismatched transplant strategies have been remarkable for a low transplant related mortality rate, but a still formidable risk of GVHD and graft rejection. In this trial, we have incorporated a combination ex-vivo T-cell depletion strategy to prevent GVHD with vigorous in vivo depletion of host (and to a lesser extent donor) T-cells to prevent graft rejection.

Patients will receive non-myeloablative conditioning with cyclophosphamide, thymoglobulin, fludarabine, and thymic irradiation, followed by a T-cell depleted PBSC infusion. Cyclosporine will be given for GVHD prophylaxis, and tapered beginning on day 35. Data from our mouse model and previous clinical trials have demonstrated that this approach can induce mixed chimerism without GVHD, with the potential for conversion of mixed chimerism to full donor hematopoiesis following donor leukocyte infusions.

ELIGIBILITY:
Inclusion Criteria:

* Disease statue: NHL, HD, or MM that are chemorefractory or relapsed; CLL that is Rai Stage III/IV, or lymphocyte doubling time of 6 months, or stage I/II that is resistant to > 2 chemotherapy regimens; AML or ALL in 1st or subsequent remission with poor prognostic features; CML in accelerated or blast phae; MDS with life-threatening cytopenias; patients who have had a previous autologous or allogeneic bone marrow or stem cell transplant; other hematologic disorders which allogeneic stem cell transplantation is appropriate where the risk of conventional transplantation is considered to be unacceptably high.
* Estimated disease-free survival of less than one year
* ECOG performance status of 0, 1, or 2
* HLA-genotypically or phenotypically matched (at A, B, DR loci) related donor

Exclusion Criteria:

* Patients who life expectancy is limited by diseases other than their hematologic malignancy.
* Cardiac Disease: symptomatic congestive hearth failure, or RVG, or ejection fraction of < 45%, active angina pectoris, or uncontrolled hypertension.
* Pulmonary Disease: severe chronic obstructive lung disease, or symptomatic restrictive lung disease, or DLCO of < 50%.
* Renal Disease: serum creatinine > 2.0 mg/dl or creatinine clearance < 50 ml/min.
* Hepatic Disease: serum bilirubin > 2.0 mg/dl or alkaline phosphatase, SGOT or SGPT > 3 times normal.
* Neurologic Disease: symptomatic leukoencephalopathy, active CNS malignancy or other neuropsychiatric abnormalities believed to preclude transplantation
* HIV or HTLV I antibody or Hepatitis B surface antigen positivity
* Uncontrolled infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the risks of severe (grade III/IV) GVHD or transplant related mortality at < 100 days following HLA-matched non-myeloablative stem cell transplantation (or following "prophylactic" DLI given for chimerism conversion). | 100 days

SECONDARY OUTCOMES:
To evaluate the incidence of acute and chronic GVHD. | indefinite
To evaluate the incidence of graft loss. | 100 days
To evaluate progression free and overall survival. | indefinite

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spitzer, M.D., Principal Investigator — Massachusetts General Hospital, Harvard University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No